CLINICAL TRIAL: NCT01418417
Title: A Randomized, Open Label, Two Treatment, Two Period, Two Sequence, Single Dose, Crossover, Bioequivalence Study of Pantoprazole Sodium 40 mg Delayed Release Tablets of Torrent Pharmaceutical Limited., India and Protonix® (Pantoprazole Sodium) 40 mg Delayed Release Tablets of Wyeth Pharmaceuticals Inc, in Healthy Human Adult Subjects, Under Fasting Conditions
Brief Title: Bioequivalence Study of Torrent Pharmaceutical Limited's Pantoprazole Sodium 40 mg Delayed Release Tablets Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Torrent Pharmaceuticals Limited (Industry)
Responsible Party: Chief Investigator, Torrent Pharmaceuticals Limited
Other Study IDs: 1200/07
Record Dates: First submitted 2011-08-10; First posted 2011-08-17 (Estimated); Last update posted 2011-08-17 (Estimated); Status verified 2011-08

CONDITIONS: Healthy

INTERVENTIONS:
Drug: Torrent's Pantoprazole Sodium Delayed - Release Tablets

SUMMARY:
Objective:

To compare the single dose bioavailability of Torrent's Pantoprazole Sodium Delayed - Release Tablets 1 × 40 mg and PROTONIX® (Pantoprazole Sodium) Delayed - Release Tablets 1 × 40 mg of Wyeth Pharmaceutical Inc. Dosing periods were separated by a washout period of at least 7 days.

Study Design:

randomized, open label, two treatment, two period, two sequence, single dose, crossover study in healthy human adult subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy human adult subjects between 18-55 years of age (inclusive), having a body mass index (BMI) between 18 and 27 kg/m2.
* Subjects who have no evidence of underlying disease during screening history and whose physical examination is performed within 21 days prior to commencement of the study.
* Subjects whose screening laboratory values are within normal limits or considered by the physician/Principal Investigator to be of no clinical significance.
* Informed consent given in written form according to section 11.3 of the protocol.
* Female Subjects:

  1. Of child bearing potential practicing an acceptable method of birth control for the duration of the study as judged by the investigator(s), such as condoms, foams, jellies, diaphragm, intrauterine device (IUD), or abstinence.
  2. Postmenopausal for at least 1 year.
  3. Surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy has been performed on the subject).

Exclusion Criteria:

* History or presence of significant:

  1. Cardiovascular, pulmonary, hepatic, renal, hematological, gastrointestinal, endocrine, immunologic, dermatologic, musculoskeletal, neurological or psychiatric disease.
  2. Alcohol dependence, alcohol abuse or drug abuse within past one year.
  3. Moderate to heavy smoking (>10 cigarettes/day) or consumption of tobacco products.
  4. History of difficulty in swallowing tablet / capsule.
  5. Clinically significant illness within 4 weeks before the start of the study
  6. Asthma, urticaria or other allergic type reactions after taking any medication.
  7. Positive urine drug screening, HIV, Hepatitis B & C tests.
  8. Any history of hypersensitivity to Pantoprazole Sodium.
  9. Existence of any surgical or medical condition, which, in the judgment of clinical investigator might interfere with the pharmacokinetics of the drug or likely to compromise the safety of the subject.
  10. Inability to communicate or co-operate with the investigator due to language problem, attitude, poor mental development / impaired cerebral function.
* Subject who has participated in any other clinical trial involving drug administration and collection of blood samples or has donated blood in the preceding 12 weeks prior to the start of the study.
* Subjects who have:

  1. Systolic blood pressure less than 90 mm of Hg or more than 150 mm of Hg.
  2. Diastolic blood pressure less than 60 mm of Hg or more than 94 mm of Hg. 3) Minor deviations (2-4 mm Hg) at check-in may be acceptable at the discretion of the physician /investigator.

  4) Pulse rate below 50/minute or above 105/minute.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult

PRIMARY OUTCOMES:
Bioequivalence based on Cmax parameter
  bioequivalence; 90% geometric confidence interval of the ratio of least-squares means of the test to reference product should be within 80.00% - 125.00% for Cmax
Bioequivalence based AUC parameter
  bioequivalence; 90% geometric confidence interval of the ratio of least-squares means of the test to reference product should be within 80.00% - 125.00% for AUC-unf, AUC(o-t).

CONTACTS AND LOCATIONS:
Locations (1):
- Lotus Labs Pvt. Ltd., Bangalore, Karnataka, India